CLINICAL TRIAL: NCT05780775
Title: Study of Lipid Balance in Adult Sickle Cell SS or SC Patients at Steady State and According to Clinical Phenotypes and During Acute Complications Acronym : "HDL2"
Brief Title: Lipid Balance in Adult Sickle Cell Patients
Acronym: HDL2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PAP_RIPH2_2021/09
Record Dates: First submitted 2022-12-12; First posted 2023-03-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease; Dyslipidemia; Complication
Keywords: Sickle cell disease; lipids; vasoocclusive crisis; priapism; pulmonary arterial hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Dyslipidemias; Vaso-Occlusive Crises; Priapism; Pulmonary Arterial Hypertension | interventions — Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HDL 2 follow up (Other): Cohort of adult sickle cell anemia (SCA) and SC sickle cell patients living in Guadeloupe and followed by SCD Reference and Competence Center of Guadeloupe.
  Interventions: Other: HDL2

INTERVENTIONS:
Other: HDL2 — to perform additional blood samples during acute phase of complications (realized between Day 1 and Day 3) in SCD patients hospitalized for vasoocclusive crisis or priapism.
  Other Names: collection of plasma and of cells.

SUMMARY:
This study aims to describe and/or searches for, in cohorts of adult sickle cell anemia (SCA) and SC sickle cell patients living in the French West Indies and followed by SCD Reference and Competence Centers: 1-lipids profiles and associations at steady state with occurrence of sickle cell disease (SCD) complications, 2-lipids profile evolution during and after prospective acute complications (vasoocclusive crises (VOC) and priapism), 3-lipids profile variation (inter /intra individuals) during 4 prospective years, 4- Genetic primary modulators of SCD complications, 5- insulin resistance (HOMA), free fatty acids and glycerol dosages, 6- lipids enzymes, lipidome and functionality of HDL in sub-groups of SCD population.

DETAILED DESCRIPTION:
* Cohorts of sickle cell disease patients including sickle cell anemia (SCA) and SC sickle cell patients living in Guadeloupe and Martinique and followed by the Sickle cell disease (SCD) Reference and Competence Centers of French West Indies.
* Lipid profile includes total cholesterol, HDL-cholesterol, non-HDL-cholesterol, LDL-cholesterol and triglycerides, apolipoprotein A-I and B.

Medical histories and prospective collection of SCD complications include retinopathy, deafness, tinnitus, osteonecrosis, leg ulcers, strokes, acute chest syndrome, VOC, priapism, pulmonary arterial hypertension (PAH) and PAH sd (echocardiography diagnosed when tricuspid regurgitant jet velocity ≥2.5 m/sec), kidney disease: chronic renal insufficiency and/or nephropathy.

* Objective 4: to describe genetic primary modulators of SCD complications: fetal hemoglobin, alpha-thalassemia, haplotypes of beta S gene.
* Objective 5 will be performed in the entire cohort at inclusion and during prospective complications (VOC, priapism).
* Objective 6 will be performed in a sub-group of 90 individuals (n=15 with VOC and n= 15 without VOC, n=15 with priapism and n=15 without priapism, n= 15 with pulmonary arterial hypertension syndrome (PAH Sd) and n=15 without PAH Sd), as well as in a subgroup of n = 15 patients prospectively experiencing VOC and n = 15 patients prospectively experiencing priapism.

A collection of plasma is performed to fulfill objective 6, as well as a collection of blood cells for later researches.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years and over
* Be affected with Sickle cell anemia or SC sickle cell
* Living in French Caribbean Islands of Guadeloupe or Martinique and followed by physicians issued from a French West Indies Sickle Cell Reference or Competence Center
* At steady state in the last month (without acute complication)
* To have given a written consent after information on the study.

Exclusion Criteria:

* Other hemoglobinopathies than sickle cell disease
* Pregnancy or lactation
* Patient under judicial protection or without freedom
* Patient not affiliated with a social security system
* Patient hospitalized for transfusion or bleeding in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
/ Lipids profiles at steady state, in sickle cell anemia and SC sickle cell adult patients, classified according to occurrence of complications. | 6 years
  Cohorts of sickle cell disease patients include sickle cell anemia (SCA) and SC sickle cell patients living in Guadeloupe and Martinique and followed by the Sickle cell disease (SCD) Reference and Competence Centers of French West Indies.
  Lipid profile includes total cholesterol, HDL-cholesterol, non-HDL-cholesterol, LDL-cholesterol and triglycerides, apolipoproteins A-I and B.
  Collection of medical histories and of prospective SCD complications include retinopathy, deafness, tinnitus, osteonecrosis, leg ulcers, strokes, acute chest syndrome, VOC, priapism, pulmonary arterial hypertension (PAH) and PAH sd (echocardiography diagnosed when tricuspid regurgitant jet velocity ≥2.5 m/sec), kidney disease: chronic renal insufficiency and/or nephropathy

SECONDARY OUTCOMES:
Kinetic study of lipids profile during hospitalized vasoocclusive crisis (VOC, with or without ACS) and Priapism, at return to steady state at first annual check-up, and one year after this last measurement | 6 years
  Past and prospective collection of previously listed SCD complications
Study of variation of lipid profile, at steady state, during a 4 years period study intra and inter individual levels. | 6 years
  total cholesterol
Study of variation of lipid profile, at steady state, during a 4 years period study intra and inter individual levels. | 6 years
  HDL-cholesterol
Study of variation of lipid profile, at steady state, during a 4 years period study intra and inter individual levels. | 6 years
  non HDL-cholesterol
Study of variation of lipid profile, at steady state, during a 4 years period study intra and inter individual levels. | 6 years
  LDL-cholesterol
Study of variation of lipid profile, at steady state, during a 4 years period study intra and inter individual levels. | 6 years
  triglycerides
Study of variation of lipid profile, at steady state, during a 4 years period study intra and inter individual levels. | 6 years
  Apolipoproteins A-I and B
Description of genetic primary modulators of SCD complications. | 6 years
  Fetal hemoglobin,
Description of genetic primary modulators of SCD complications. | 6 years
  alpha-thalassemia,
Description of genetic primary modulators of SCD complications. | 6 years
  haplotypes of beta S gene
Dosages of Insulin resistance (HOMA), | 6 years
  Plasmatic insulinemia and glycemia (HOMA) will be performed in the entire cohort at inclusion and during prospective complications (VOC, priapism); lipids dosages
free fatty acids | 6 years
  kinetic study of free fatty acids at inclusion and during prospective complications (VOC, priapism);
plasmatic glycerol. | 6 years
  Kinetic study of plasmatic at inclusion and during prospective complications (VOC, priapism);
Dosages of lipids enzymes, lipidome and functionality of HDL at steady state | 6 years
  The dosages of CETP (Cholesteryl Ester Transfer Protein) enzymes activities
Dosages of lipids enzymes, lipidome and functionality of HDL at steady state | 6 years
  The dosages of L-CAT (Lécithine Cholestérol Acyl Transférase) enzymes activities
Dosages of lipids enzymes, lipidome and functionality of HDL at steady state | 6 years
  The dosages of HDL lipidome,
Dosages of lipids enzymes, lipidome and functionality of HDL at steady state | 6 years
  The dosages of HDL functionality,
Dosages of lipids enzymes, lipidome and functionality of HDL at steady state | 6 years
  The dosages of free fatty acid
Dosages of lipids enzymes, lipidome and functionality of HDL at steady state | 6 years
  The dosages of glycerol

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure LALANNE-MISTRIH, Principal Investigator — : University Hospital of Guadeloupe - Department of Nutrition
Locations (1):
- Unité Transversale de la Drépanocytose, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No